CLINICAL TRIAL: NCT06924060
Title: EFFECT OS RESISTANCE TRAINING VOLUME WITH INERTIAL FLYWHEEL ON MUSCLE ADAPTATIONS IN UNTRAINED MEN: A RANDOMIZED CLINICAL TRIAL
Brief Title: EFFECT OF RESISTANCE TRAINING VOLUME WITH INERTIAL FLYWHEEL ON MUSCLE ADAPTATIONS IN UNTRAINED MEN
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Vicosa (Other)
Responsible Party: Principal Investigator, Suene Franciele Nunes Chaves, PhD Student, Federal University of Vicosa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81740024.5.0000.5153
Record Dates: First submitted 2025-03-31; First posted 2025-04-11 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Resistance Training; Eccentric Exercise Training
Keywords: randomized clinical trial; flywheel resistance training; hypertrophy; maximum voluntary isometric contraction
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Hidden and opaque envelope technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2 sets group (Experimental): Group that will perform two sets of each exercise developed during the intervention. The other training variables will be identical (repetitions, moment of inertia, rest intervals between sets and repetitions, rest intervals between workouts, training frequency, number and order of exercises).
  Interventions: Behavioral: Flywheel Resistance Training with two sets
- 4 sets group (Experimental): Group that will perform four sets of each exercise developed during the intervention. The other training variables will be identical (repetitions, moment of inertia, rest intervals between sets and repetitions, rest intervals between workouts, training frequency, number and order of exercises).
  Interventions: Behavioral: Flywheel Resistance Training with four sets
- 6 sets arm (Experimental): Group that will perform six sets of each exercise developed during the intervention. The other training variables will be identical (repetitions, moment of inertia, rest intervals between sets and repetitions, rest intervals between workouts, training frequency, number and order of exercises).
  Interventions: Behavioral: Flywheel Resistance Training with six sets

INTERVENTIONS:
Behavioral: Flywheel Resistance Training with two sets — For each training session, 4 generic exercises will be performed, involving small and large muscle groups (leg extension, leg flexion, biceps curl, triceps french press). They will perform 2 sets of 8 repetitions, with a 2-minute break between exercises and sets. They will perform these exercises at a high intensity (always 10 on the OMNI-RES Scale).
  Other Names: Flywheel Inertial Training; Eccentric Training
  Arms: 2 sets group
Behavioral: Flywheel Resistance Training with four sets — For each training session, 4 generic exercises will be performed, involving small and large muscle groups (leg extension, leg flexion, biceps curl, triceps french press). They will perform 4 sets of 8 repetitions, with a 2-minute break between exercises and sets. They will perform these exercises at a high intensity (always 10 on the OMNI-RES Scale).
  Other Names: Flywheel Inertial Training; Eccentric Training
  Arms: 4 sets group
Behavioral: Flywheel Resistance Training with six sets — For each training session, 4 generic exercises will be performed, involving small and large muscle groups (leg extension, leg flexion, biceps curl, triceps french press). They will perform 6 sets of 8 repetitions, with a 2-minute break between exercises and sets. They will perform these exercises at a high intensity (always 10 on the OMNI-RES Scale).
  Other Names: Flywheel Inertial Training; Eccentric Training
  Arms: 6 sets arm

SUMMARY:
Muscular strength is essential for health and quality of life, impacting body composition, balance, locomotion, functional independence, and mental health. Resistance training (RT) is the primary way to increase strength and muscle hypertrophy. Traditionally, RT programs rely on gravity, which can limit muscle activation, especially during the eccentric phase of movement. To improve outcomes, it is important to include methods that intensify muscle work during this phase.

Flywheel resistance Training (FWRT) was developed to increase overload during the eccentric phase by harnessing the energy generated during the concentric phase and applying it to the eccentric phase. This type of training has shown positive results in several studies, improving strength, hypertrophy, jump performance, aerobic endurance, agility, and running economy.

However, there are still no studies that define how the variables of FWRT should be effectively prescribed. Properly adjusting these variables can optimize muscle adaptations and improve physical fitness and health indices. Therefore, in this study, the number of sets will be evaluated to investigate whether a higher number of sets can lead to greater muscle adaptations.

DETAILED DESCRIPTION:
Thirty young men will be randomly assigned to three groups: 2 sets, 3 sets, and 4 sets of Flywheel Resistance Training (FWRT). The interventions will take place at the Department of Physical Education at the Federal University of Vicosa, with all sessions supervised by certified physical education professionals. Follow-up will be conducted through WhatsApp messages and phone calls. All groups will train twice a week for eight weeks. Participants from all experimental groups will perform FWRT on a multi-leg isoinertial machine targeting both upper and lower body muscles. Each session will include 4 exercises, performed for 8 repetitions, with a 2-minute rest between sets and exercises. Training progression will be adjusted based on the participant's ability to exceed the suggested maximum repetitions with the same mobilized weight. The exercises will target various muscle groups, including leg extensions, leg curls, bicep curls, and triceps french press.

Participants will be evaluated at two points during the training program: pre-intervention and post-intervention. Muscle strength of the upper and lower limbs will be assessed through one-repetition maximum (1RM) tests on a knee extension or elbow flexion machine and through maximum voluntary isometric contraction (MVIC), evaluated with a load cell. The muscle thickness of the knee extensors and elbow flexors will be measured using a B-mode ultrasound. Load control will be monitored through the following scales: Total Quality of Recovery (TQR) and Visual Analog Scale for Delayed Onset Muscle Soreness (VAS-DOM), and after each set, by the Subjective Perception of Effort (OMNI-RES). To ensure adequate protein intake, at the end of each training session, participants will receive a dose of Whey Protein, based on data collected from their initial food recall and determined by a nutritionist. Anthropometric evaluation will include the measurement of: a) body mass using an electronic/digital scale with 100g resolution , and b) height using a millimetric stadiometer. The procedures used for body mass and height measurement will follow the protocols based on the measurement standards of the International Society for the Advancement of Anthropometry.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported levels of speaking, writing and understanding Portuguese;
2. Availability to participate in the research (initial meeting, initial and final tests, data collection);
3. Have not been performing traditional resistance exercises for at least 6 months (untrained subjects);
4. Have no previous experience with inertial flywheel devices;
5. Answer no to all questions on the Physical Activity Risk Questionnaire - PAR-Q;
6. Have no medical contraindication of any kind.

Exclusion Criteria:

1. Have a history of recent osteomyoarticular injury;
2. Have uncontrolled chronic diseases;
3. Surgical procedures scheduled during interventions;
4. Do not have the flexibility to adapt their diet to the guidelines offered during collection;
5. Use medications or supplements that may interfere with the result, acting as an intervening variable.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Maximum isometric voluntary contraction (upper extremities) | Baseline and after eight weeks
  To evaluate the Maximum isometric voluntary contraction (MIVC) of the upper extremities, a load cell or extensometric cell with a sampling frequency of 1000 Hz will be used.
Maximum isometric voluntary contraction (lower extremities) | Baseline and after eight weeks
  To evaluate the Maximum isometric voluntary contraction (MIVC) of the lower extremities, a load cell or extensometric cell with a sampling frequency of 1000 Hz will be used.
1 RM test (elbow flexors) | Baseline and after eight weeks
  To perform the one repetition maximum (1RM) test, the load cell will be placed on a Cross Over machine (Scorpions Fitness, Brazil), so that one of its ends is fixed by means of a chain to the lower part of a stirrup-type handle and the other end is fixed to the steel cable, which is subjected to traction when the machine's lever arm is moved. Before performing the test, the device will be adjusted so that the subject's elbow is at a 90° flexion angle.
1 RM test (knee extension) | Baseline and after eight weeks
  To perform the one repetition maximum test (1RM), the knee extension exercise or elbown flexion will be used on a BH fitness® Nevada Pro-t extension machine. To perform the test, the volunteer will be asked to extend the knee to form an angle of approximately 180° (final position) and return to the initial position.
Muscle power (upper extremities) | Baseline and after eight weeks
  The evaluation of power elbow flexors will be assessed using the same machine used to assess 1RM. The load for assessing power should be used, obtained from the percentage value of 1RM (40%, 60% and 80% of 1RM), so that the subject performs the elbow flexion movement (concentric phase of the movement) at the highest possible speed. The return of the elbow to the initial position will be performed in a controlled manner, with a pause of one to two seconds, to prevent the effect of the accumulated elastic force from interfering with the next execution. A linear position transducer or Encoder will be used, with a sampling frequency of 1000 Hertz to determine the power values. Through this instrument it will be possible to obtain information on average muscle power (MMP) and peak muscle power (PP).
Muscle power (lower extremities) | Baseline and after eight weeks
  The evaluation of lower limb muscle power will be performed using the same knee extension machine used in the exercise sessions, starting from the same initial position (90º of kneeling flexion) and reaching the same final position (180º of knee extension) as the test of 1RM. The load for assessing power should be used, obtained from the percentage value of 1RM (40%, 60% and 80% of 1RM), so that the subject performs the knee extension movement (concentric phase of the movement) at the highest possible speed. The return of the knee to the initial position will be performed in a controlled manner, with a pause of one to two seconds, to prevent the effect of the accumulated elastic force from interfering with the next execution. A linear position transducer or Encoder will be used, with a sampling frequency of 1000 Hertz.
Muscle adaptations | Baseline and after eight weeks
  The muscle thickness of the knee extensors and elbow flexors will be measured using a B-mode ultrasound. Image acquisition will be performed by an experienced and previously trained researcher. The image will be considered suitable for analysis when the muscle-bone and subcutaneous adipose tissue-muscle interfaces are identified. The image will then be saved and analyzed in Image-J by the same experienced evaluator.

SECONDARY OUTCOMES:
Delayed Onset Muscle Soreness | Before each training session during the 8 weeks of intervention
  To assess the history of Delayed Onset Muscle Soreness, the Visual Analog Scale for Delayed Onset Muscle Soreness (VAS-DOM) will be used to identify whether there are changes throughout the intervention for this variable, that is, whether the volunteer gets used to the intervention and feels less pain throughout the sessions.
Subjective Perception of Effort | Before each training session during the 8 weeks of intervention
  To assess the subjective perception of effort, the Subjective Perception of Effort (OMINI-RES) scale will be used, in order to identify whether there are changes throughout the intervention for this variable, that is, whether the volunteer gets used to the intervention and feels a lower perception of effort throughout the sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo C Moreira, PhD supervisor, Study Director — Federal University of Viçosa
Locations (1):
- Federal University at Viçosa, Viçosa, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No